CLINICAL TRIAL: NCT05039034
Title: Screening and Management of High-risk Populations of Stroke in Dehui City
Acronym: SAMHPSDC
Status: Completed | Type: Observational
Sponsor: Yi Yang (Other)
Collaborators: Dehui People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: SMDC
Record Dates: First submitted 2021-08-30; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Cerebrovascular Accident; Stroke; Hypertension; Diabetes Mellitus; Dyslipidemias
Keywords: Stroke/epidemiology; Stroke/prevention and control; Risk Factors; Cognition; Surveys and Questionnaires
MeSH Terms: conditions — Stroke; Hypertension; Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Low-risk Group: Low-risk Group is defined as the population with <3 risk factors (hypertension, dyslipidemia or dyslipoproteinemia, diabetic mellitus, atrial fibrillation or valvular heart disease, smoking, lack of exercise or light manual labor, overweight or obesity and family history of stroke), but without chronic disease (hypertension, diabetic mellitus, atrial fibrillation or valvular heart disease).
  Interventions: Other: Advice according to primary prevention guidelines on stroke of China
- Mediate-risk Group: Mediate-risk Group is defined as the population with <3 risk factors (hypertension, dyslipidemia or dyslipoproteinemia, diabetic mellitus, atrial fibrillation or valvular heart disease, smoking, lack of exercise or light manual labor, overweight or obesity and family history of stroke), but meanwhile suffer from chronic disease (hypertension, diabetic mellitus, atrial fibrillation or valvular heart disease).
  Interventions: Other: Advice according to primary prevention guidelines on stroke of China
- High-risk Group: High-risk Group is defined as the population with ≥3 risk factors (hypertension, dyslipidemia or dyslipoproteinemia, diabetic mellitus, atrial fibrillation or valvular heart disease, smoking, lack of exercise or light manual labor, overweight or obesity and family history of stroke), or population with history of stroke or/and transient ischemic attack.
  Interventions: Other: Advice according to primary prevention guidelines on stroke of China

INTERVENTIONS:
Other: Advice according to primary prevention guidelines on stroke of China

SUMMARY:
This epidemiological survey is to analyze the prevalence rate of stroke and exposure rate of risk factors in sampling population aged 40 years and over (born before December 31,1975) in Dehui City, to provide scientific basis for pertinent prevention and control of stroke in Jilin Province, and to provide valuable data for the high-risk groups to carry out regular follow-up and standardized management.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years and over in Dehui City
* Willing to participate in the study and follow-up visits
* Signed an informed consent

Exclusion Criteria:

* Life expectancy<3 years
* Unwilling to participate in the study and follow-up visits
* Living away from Dehui City over 6 months
* Unable to cooperate with examination and questionnaire due to mental disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Target population aged 40 years and over (born before December 31,1975) was selected from Dehui City by means of group sampling.
Sampling Method: Probability Sample
Enrollment: 4100 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Prevalence rate of stroke | 4 months
  The proportion of stroke in the general population.
Prevalence rate of hypertension | 4 months
  The proportion of hypertension in the general population.
Prevalence rate of diabetes mellitus | 4 months
  The proportion of diabetes mellitus in the general population.
Prevalence rate of dyslipidemia | 4 months
  The proportion of dyslipidemia in the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, M.D. Ph.D., Study Chair — The First Hospital of Jilin University; Ying-Qi Xing, M.D. Ph.D., Study Director — The First Hospital of Jilin University; Zhen-Ni Guo, M.D., Study Director — The First Hospital of Jilin University; Fu-Liang Zhang, M.D., Principal Investigator — The First Hospital of Jilin University; Hao-Yuan Liu, M.D., Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China